CLINICAL TRIAL: NCT04740931
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Macular Edema Secondary to Central Retinal or Hemiretinal Vein Occlusion
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab in Participants With Macular Edema Secondary to Central Retinal or Hemiretinal Vein Occlusion
Acronym: COMINO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR41986; 2020-000441-13 (EudraCT Number)
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion; Hemiretinal Vein Occlusion
Keywords: CRVO; HRVO
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — faricimab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) (Experimental): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm A will receive faricimab 6 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants will receive faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure will be administered during study visits at which no faricimab treatment is administered (according to the PTI dosing regimen).
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) (Active Comparator): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm B will receive aflibercept 2 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants will receive faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure will be administered during study visits at which no faricimab treatment is administered (according to the PTI dosing regimen).
  Interventions: Drug: Faricimab; Drug: Aflibercept; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by intravitreal (IVT) injection as specified in each treatment arm.
  Other Names: VABYSMO®; faricimab-svoa; RG7716; RO6867461
Drug: Aflibercept — Aflibercept 2 mg will be administered by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
  Other Names: Eylea
  Arms: Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Procedure: Sham Procedure — The sham is a procedure that mimics an IVT injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. It will be administered to participants in both treatments arms at applicable visits to maintain masking.

SUMMARY:
This is a Phase III, multicenter, randomized, double-masked, active comparator-controlled, parallel-group study evaluating the efficacy, safety, and pharmacokinetics of faricimab administered by intravitreal (IVT) injection at 4-week intervals until Week 24, followed by a double-masked period of study without active control to evaluate faricimab administered according to a personalized treatment interval (PTI) dosing regimen in patients with macular edema due to central retinal vein occlusion (CRVO) or hemiretinal vein occlusion (HRVO).

ELIGIBILITY:
Inclusion Criteria:

* Foveal center-involved macular edema due to central retinal vein occlusion (CRVO) or hemiretinal vein occlusion (HRVO), diagnosed no longer than 4 months prior to the screening visit
* Best-corrected visual acuity (BCVA) of 73 to 19 letters, inclusive (20/40 to 20/400 approximate Snellen equivalent)
* Sufficiently clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm diagnosis
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs during the treatment period and for 3 months after the final dose of study treatment

Exclusion Criteria:

* Any major illness or major surgical procedure within 1 month before screening
* Uncontrolled blood pressure
* Stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to Day 1
* Pregnant or breastfeeding, or intending to become pregnant during the study

Ocular Exclusion Criteria for Study Eye:

* History of previous episodes of macular edema due to RVO or persistent macular edema due to RVO diagnosed more than 4 months before screening
* Any current ocular condition which, in the opinion of the investigator, is currently causing or could be expected to contribute to irreversible vision loss due to a cause other than macular edema due to RVO in the study eye (e.g., ischemic maculopathy, Irvine-Gass syndrome, foveal atrophy, foveal fibrosis, pigment abnormalities, dense subfoveal hard exudates, or other non-retinal conditions)
* Macular laser (focal/grid) in the study eye at any time prior to Day 1
* Panretinal photocoagulation in the study eye within 3 months prior to Day 1 or anticipated within 3 months of study start on Day 1
* Any prior or current treatment for macular edema; macular neovascularization, including diabetic macular edema (DME) and neovascular age-related macular degeneration (nAMD); and vitreomacular-interface abnormalities, including, but not restricted to, IVT treatment with anti-VEGF, steroids, tissue plasminogen activator, ocriplasmin, C3F8, air or periocular injection
* Any prior intervention with verteporfin photodynamic therapy, diode laser, transpupillary thermotherapy, or vitreo-retinal surgery including sheathotomy
* Any prior steroid implant use including dexamethasone intravitreal implant (Ozurdex) and fluocinolone acetonide intravitreal implant (Iluvien)

Ocular Exclusion Criteria for Both Eyes:

* Prior IVT administration of faricimab in either eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active periocular, ocular or intraocular inflammation or infection (including suspected) in either eye on Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (194):
- United States (57):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Oakland, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - West Coast Retina Medical Group, San Francisco, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Advanced Research, Deerfield Beach, Florida
  - Rand Eye, Deerfield Beach, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Northwestern Medical Group/Northwestern University, Chicago, Illinois
  - Retina Associated Ltd, Elmhurst, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Retina Center, Springfield, Illinois
  - Retina Associates, Lenexa, Kansas
  - Johns Hopkins Med; Wilmer Eye Inst, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC.; DBA Retina Consultants of Minnesota, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - Retina Assoc of Western NY, Rochester, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Northwest, Portland, Oregon
  - Cascade Medical Research Institute LLC, Springfield, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Argentina (9):
  - Fundacion Zambrano, CABA
  - Centro Oftalmológico Dr. Charles S.A., Capital Federal
  - Oftalmos, Capital Federal
  - Hospital Italiano; Ophtalmology, Capital Federal
  - Buenos Aires Mácula, Ciudad Autonoma Buenos Aires
  - Oftar, Mendoza
  - Centro Oftalmólogos Especialistas, Rosario
  - Grupo Laser Vision, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Australia (7):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Save Sight Institute, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Austria (2):
  - LKH-Univ.Klinikum Graz; Universitäts-Augenklinik, Graz
  - Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna
- Brazil (5):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Universidade Federal de Sao Paulo - UNIFESP*X; Oftalmologia, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- China (15):
  - Beijing Hospital of Ministry of Health, Beijing
  - The Second Hospital of Jilin University, Changchun
  - West China Hospital, Sichuan University, Chengdu
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - Shanghai Tenth People's Hospital, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - He Eye Specialist Shenyang Hospital, Shenyang
  - The University of Hong Kong-Shenzhen Hospital; Local Ethic Committee, Shenzhen
  - Tianjin Eye Hospital, Tianjin
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Renmin Hospital of Wuhan University, Wuhan
  - Henan Provincial Eye Hosptial, Zhengzhou
- Czechia (2):
  - General Teaching Hospital Prague; Ophthalmology clinic, Prague
  - AXON Clinical, Prague
- France (4):
  - Chi De Creteil; Ophtalmologie, Créteil
  - Hopital Lariboisiere; Ophtalmologie, Paris
  - Centre Ophtalmologique; Imagerie et laser, Paris
  - Centres Ophtalmologique St Exupéry; Ophtalmologie, Saint-Cyr-sur-Loire
- Germany (3):
  - Internationale Innovative Ophthalmochirurgie GbR; c/o Makula-Netzhaut-Zentrum Breyer Kaymak Klabe, Düsseldorf-Oberkassel
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH; Augenklinik, Ludwigshafen
- Hong Kong (2):
  - Queen Mary Hospital; Department of Ophthalmology, Hong Kong
  - Hong Kong Eye Hospital; CUHK Eye Centre, Mong Kok
- Hungary (5):
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecen
  - Szegedi Tudományegyetem ÁOK; Department of Ophtalmology, Szeged
  - Zala Megyei Kórház; SZEMESZET, Zalaegerszeg
- Israel (5):
  - Rambam Medical Center; Opthalmology, Haifa
  - Hadassah MC; Ophtalmology, Jerusalem
  - Rabin MC; Ophtalmology, Petah Tikva
  - Kaplan Medical Center; Ophtalmology, Rehovot
  - Tel Aviv Sourasky MC; Ophtalmology, Tel Aviv
- Italy (2):
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
- Japan (20):
  - Sugita Eye Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Hyogo Medical University Hospital, Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Mie University Hospital, Mie
  - Fukushima Medical University Hospital, Miyagi
  - Shinshu University Hospital, Nagano
  - Osaka Metropolitan University Hospital, Osaka
  - Kansai Medical University Medical Center, Osaka
  - Tokyo Women's Medical University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Poland (17):
  - Szpital sw. Lukasza, Bielsko-Biala
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Specjalistyczny O?rodek Okulistyczny Oculomedica, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Dobry Wzrok Sp Z O O, Gda?sk
  - Optimum Profesorskie Centrum Okulistyki, Gda?sk
  - Poradnia Okulistyczna i Salon Optyczny w Gliwicach- PRYZMAT, Gliwice
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne Dietla 19 Sp. Z O.O., Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - MT Medic Krosno, Krosno
  - O?rodek Chirurgii Oka Prof. Zagórskiego Na??czów, Na??czów
  - Centrum Medyczne Pulawska SP. z o.o., Piaseczno
  - Lens Clinic, Rybnik
  - Caminomed, Tarnowskie Góry
  - Centrum Zdrowia MDM, Warsaw
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Portugal (3):
  - Centro Hospitalar E Universitário de Coimbra EPE - Serviço Oftalmologia; Serviço Oftalmologia, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Hospital de Santa Maria; Servico de Oftalmologia, Lisbon
- Russia (5):
  - Clinic Optimed, Ufa, Bashkortostan Republic
  - Intersec Research and Technology Complex ?Eye Microsurgery? n.a. S.N. Fyodorov; Cheboksary Branch, Cheboksary, Mariy-El Republic
  - FSBI ?Scientific Research Institute of Eye Diseases? of Russian Academy of medical Sciences, Moscow, Moscow Oblast
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg, Sankt-Peterburg
  - 1 Saint-Petersburg St. Med. University named after academician I.P.Pavlov; Chair of ophathalmology, Saint Petersburg, Sankt-Peterburg
- Singapore (2):
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital; Ophthalmology Department, Singapore
- South Korea (8):
  - Pusan National University Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (8):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra; Servicio de oftalmologia, Pamplona, Navarre
  - Centro de Oftalmologia Barraquer; Servicio Oftalmologia, Barcelona
  - Hospital Clinic de Barcelona; Consultas Externas Oftalmologia, Barcelona
  - Hospital de Santa Creu I Sant Pau; Servicio de Oftalmologia, Barcelona
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- Taiwan (3):
  - Changhua Christian Hospital; Department of Ophthalmology, Changhua
  - Taipei Veterans General Hospital; Ophthalmology, Taipei
  - Chang Gung Medical Foundation - Linkou; Ophthalmology, Taoyuan District
- United Kingdom (10):
  - Belfast Health and Social Care Trust, ROYAL VICTORIA HOSPITAL, Belfast
  - Birmingham Midland Eye Centre, Birmingham
  - Opthalmology Research Office, Bradford
  - Bristol Eye Hospital;Retinal Treatment and Research Unit, Bristol
  - University Hospital of Wales, Cardiff
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital; St Paul's Clinical Eye Research Centre, Liverpool
  - Central Middlesex Hospital, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Danzig CJ, Dinah C, Ghanchi F, Hattenbach LO, Khanani AM, Lai TYY, Shimura M, Abreu F, Arrisi P, Liu Y, Paris LP, Retiere AC, Willis JR, Schlottmann PG; BALATON and COMINO Investigators. Faricimab Treat-and-Extend Dosing for Macular Edema Due to Retinal Vein Occlusion: 72-Week Results from the BALATON and COMINO Trials. Ophthalmol Retina. 2025 Sep;9(9):848-859. doi: 10.1016/j.oret.2025.03.005. Epub 2025 Mar 17. PMID 40107501
- [Derived] Tadayoni R, Paris LP, Danzig CJ, Abreu F, Khanani AM, Brittain C, Lai TYY, Haskova Z, Sakamoto T, Kotecha A, Schlottmann PG, Liu Y, Seres A, Retiere AC, Willis JR, Yoon YH; BALATON and COMINO Investigators. Efficacy and Safety of Faricimab for Macular Edema due to Retinal Vein Occlusion: 24-Week Results from the BALATON and COMINO Trials. Ophthalmology. 2024 Aug;131(8):950-960. doi: 10.1016/j.ophtha.2024.01.029. Epub 2024 Jan 26. PMID 38280653

RESULTS

PARTICIPANT FLOW:
Period: Part 1 (Baseline up to Week 24)
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Started (Intent-to-Treat (ITT) Population) | 366 | 363
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 365 | 361
Completed (Completed Part 1) | 360 | 353
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Death | 1 | 2
Not completed — Non-compliance with study drug | 2 | 0
Not completed — Reason Not Specified | 2 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Part 2 (Week 24 to Week 72)
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Started | 360 | 353
Completed | 333 | 323
Not Completed | 27 | 30
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 3 | 9
Not completed — Adverse Event | 5 | 5
Not completed — Death | 4 | 1
Not completed — Other | 1 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Non-compliance with study drug | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population: All global participants who were randomized in the study, according to the assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) | Total
Number analyzed (Participants) | 366 | 363 | 729
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (13.1) | 64.7 (13.3) | 65.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 163 | 336
  Male | 193 | 200 | 393
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 66 | 73 | 139
  Not Hispanic or Latino | 286 | 283 | 569
  Unknown or Not Reported | 14 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 89 | 88 | 177
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 13 | 23
  White | 243 | 253 | 496
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 21 | 5 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Rest of World | 187 | 187 | 374
  USA and Canada | 95 | 93 | 188
  Asia | 84 | 83 | 167
Number of Participants by the Eye (Left or Right) Chosen as the Study Eye [Count of Participants; unit: Participants]
  Left Eye | 180 | 181 | 361
  Right Eye | 186 | 182 | 368
Best Corrected Visual Acuity (BCVA) Letter Score in the Study Eye [Mean (Standard Deviation); unit: ETDRS Letters] | 50.25 (16.25) | 50.71 (16.34) | 50.48 (16.29)
Number of Participants by the BCVA Letter Score Categories in the Study Eye [Count of Participants; unit: Participants]
  ≤34 Letters (20/200 or Worse) | 79 | 80 | 159
  >34 Letters to <55 Letters | 106 | 105 | 211
  ≥55 Letters (20/80 or Better) | 181 | 178 | 359

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye at Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The Mixed Model of Repeated Measures (MMRM) analysis included the categorical covariates of treatment arm, visit, visit-by-treatment arm interaction, baseline BCVA (continuous), and randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)] as fixed effects. An unstructured covariance structure was used. Missing data were implicitly imputed by MMRM model assuming missing at random. Treatment policy strategy (i.e., all observed values used) was applied to all intercurrent events (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). 95% CI is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Groups:
- Arm A: Faricimab Q4W (Part 1): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm A will receive faricimab 6 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
- Arm B: Aflibercept Q4W (Part 1): In Part 1 (Day 1 through Week 24), participants randomly assigned to Arm B will receive aflibercept 2 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections).
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
ETDRS Letters | 16.9 [15.4 to 18.3] | 17.3 [15.9 to 18.8]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); The null hypothesis, H0: μ(faricimab) - μ(aflibercept) ≤-4 letters; the alternative hypothesis, Ha: μ(faricimab) - μ(aflibercept) >-4 letters. The final sample size provided >90% power for the non-inferiority assessment (at a one-sided 0.02485 significance level); Test type: Non-Inferiority — If the lower bound of a two-sided 95% confidence interval (CI) for the difference in adjusted means of the two treatments (faricimab minus aflibercept) is greater than -4 letters (the non-inferiority margin), then faricimab is considered non-inferior to aflibercept; Difference in Adjusted Means = -0.4, 95% CI 2-sided [-2.5 to 1.6], Standard Error of Mean 1.04 — The treatment difference in adjusted means of change from baseline BCVA is the calculated difference of Arm A: Faricimab and Arm B: Aflibercept. MMRM adjustments are listed in the outcome measure description
Statistical Analysis 2: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); The final sample size provided >80% power for a 3.5-letter superiority assessment of faricimab over aflibercept (at a two-sided 0.0497 significance level); Test type: Superiority; p = 0.6715, Mixed Model of Repeated Measures — Tested at a two-sided p<0.0497 significance level; Difference in Adjusted Means = -0.4, 95% CI 2-sided [-2.5 to 1.6], Standard Error of Mean 1.04 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Part 1: Change From Baseline in BCVA in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
ETDRS Letters
  Week 4 | 13.5 [12.5 to 14.6] | 14.3 [13.2 to 15.4]
  Week 8 | 15.5 [14.4 to 16.7] | 16.5 [15.3 to 17.7]
  Week 12 | 16.9 [15.7 to 18.2] | 17.1 [15.8 to 18.4]
  Week 16 | 16.8 [15.4 to 18.1] | 17.5 [16.2 to 18.9]
  Week 20 | 17.0 [15.6 to 18.3] | 17.2 [15.8 to 18.5]
  Week 24 | 16.9 [15.4 to 18.3] | 17.3 [15.9 to 18.8]

3. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: From Baseline through Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants | 56.6 [51.7 to 61.5] | 58.1 [53.3 to 62.9]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); Test type: Other; Difference in CMH Weighted Percentage = -1.5, 95% CI 2-sided [-8.4 to 5.3]

4. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 41.5 [36.7 to 46.3] | 45.4 [40.7 to 50.2]
  Week 8 | 51.1 [46.3 to 55.9] | 53.7 [48.9 to 58.5]
  Week 12 | 54.6 [49.8 to 59.4] | 55.1 [50.3 to 59.9]
  Week 16 | 57.7 [52.8 to 62.5] | 59.5 [54.7 to 64.3]
  Week 20 | 56.6 [51.7 to 61.4] | 57.8 [53.0 to 62.6]
  Week 24 | 56.6 [51.7 to 61.5] | 58.1 [53.3 to 62.9]

5. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 60.9 [56.0 to 65.8] | 62.3 [57.6 to 66.9]
  Week 8 | 69.1 [64.5 to 73.7] | 72.8 [68.3 to 77.2]
  Week 12 | 73.2 [68.8 to 77.7] | 74.7 [70.3 to 79.0]
  Week 16 | 73.5 [69.1 to 78.0] | 75.8 [71.4 to 80.1]
  Week 20 | 72.4 [68.0 to 76.9] | 74.1 [69.7 to 78.5]
  Week 24 | 72.2 [67.7 to 76.6] | 73.3 [68.8 to 77.7]

6. Secondary Outcome: Part 1: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 83.1 [79.3 to 86.9] | 83.5 [79.7 to 87.2]
  Week 8 | 85.2 [81.7 to 88.8] | 86.8 [83.3 to 90.2]
  Week 12 | 87.4 [84.1 to 90.8] | 87.1 [83.7 to 90.5]
  Week 16 | 86.3 [82.9 to 89.8] | 88.7 [85.5 to 92.0]
  Week 20 | 84.1 [80.5 to 87.8] | 86.5 [83.0 to 90.0]
  Week 24 | 85.3 [81.8 to 88.8] | 84.6 [80.9 to 88.2]

7. Secondary Outcome: Part 1: Percentage of Participants Gaining >0 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 92.1 [89.4 to 94.8] | 95.6 [93.5 to 97.7]
  Week 8 | 92.1 [89.4 to 94.8] | 94.8 [92.5 to 97.0]
  Week 12 | 93.2 [90.6 to 95.7] | 92.6 [89.9 to 95.2]
  Week 16 | 92.6 [90.0 to 95.3] | 92.0 [89.3 to 94.8]
  Week 20 | 90.5 [87.5 to 93.4] | 91.4 [88.6 to 94.3]
  Week 24 | 90.5 [87.5 to 93.4] | 89.2 [86.1 to 92.4]

8. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 98.4 [97.1 to 99.7] | 98.9 [97.8 to 100.0]
  Week 8 | 98.1 [96.7 to 99.5] | 98.1 [96.7 to 99.5]
  Week 12 | 98.6 [97.5 to 99.8] | 97.5 [95.9 to 99.1]
  Week 16 | 97.3 [95.6 to 98.9] | 97.0 [95.2 to 98.7]
  Week 20 | 97.0 [95.3 to 98.7] | 96.7 [94.9 to 98.5]
  Week 24 | 96.2 [94.3 to 98.1] | 96.7 [94.9 to 98.5]

9. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 98.1 [96.7 to 99.5] | 98.6 [97.4 to 99.8]
  Week 8 | 97.5 [96.0 to 99.1] | 97.5 [95.9 to 99.1]
  Week 12 | 97.8 [96.3 to 99.3] | 97.0 [95.2 to 98.7]
  Week 16 | 95.9 [93.9 to 97.9] | 96.1 [94.2 to 98.1]
  Week 20 | 96.7 [94.9 to 98.5] | 96.1 [94.2 to 98.1]
  Week 24 | 95.1 [92.9 to 97.3] | 95.9 [93.8 to 97.9]

10. Secondary Outcome: Part 1: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 97.0 [95.3 to 98.7] | 98.1 [96.7 to 99.5]
  Week 8 | 96.2 [94.2 to 98.1] | 96.4 [94.5 to 98.3]
  Week 12 | 95.9 [93.9 to 97.9] | 96.1 [94.2 to 98.1]
  Week 16 | 95.4 [93.2 to 97.5] | 94.8 [92.5 to 97.0]
  Week 20 | 94.8 [92.6 to 97.1] | 93.9 [91.5 to 96.4]
  Week 24 | 94.0 [91.6 to 96.4] | 93.7 [91.2 to 96.1]

11. Secondary Outcome: Part 1: Percentage of Participants Achieving ≥84 Letters in BCVA (20/20 Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 6.0 [3.6 to 8.4] | 4.7 [2.6 to 6.8]
  Week 8 | 8.7 [5.9 to 11.5] | 10.2 [7.2 to 13.2]
  Week 12 | 10.9 [7.8 to 14.0] | 11.9 [8.7 to 15.0]
  Week 16 | 11.5 [8.4 to 14.6] | 14.1 [10.7 to 17.5]
  Week 20 | 14.2 [10.9 to 17.6] | 14.9 [11.4 to 18.3]
  Week 24 | 14.5 [11.0 to 17.9] | 15.2 [11.7 to 18.7]

12. Secondary Outcome: Part 1: Percentage of Participants Achieving ≥69 Letters in BCVA (20/40 or Better Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 45.0 [41.0 to 49.1] | 46.1 [41.9 to 50.2]
  Week 8 | 48.6 [44.3 to 52.8] | 54.6 [50.5 to 58.7]
  Week 12 | 54.9 [50.8 to 58.9] | 55.7 [51.4 to 60.0]
  Week 16 | 54.9 [50.6 to 59.1] | 59.3 [55.2 to 63.4]
  Week 20 | 54.1 [49.7 to 58.4] | 57.6 [53.4 to 61.8]
  Week 24 | 55.7 [51.3 to 60.0] | 59.0 [54.5 to 63.4]

13. Secondary Outcome: Part 1: Percentage of Participants With ≤38 Letters in BCVA (20/200 or Worse Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 24
Description: Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by baseline BCVA (>38 and ≤38 letters) and region (U.S. and Canada, Asia, and rest of the world). All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 10.0 [7.3 to 12.8] | 8.6 [6.1 to 11.1]
  Week 8 | 8.2 [5.5 to 10.8] | 7.0 [4.6 to 9.4]
  Week 12 | 7.3 [4.9 to 9.8] | 6.4 [4.0 to 8.8]
  Week 16 | 7.8 [5.3 to 10.4] | 6.2 [3.8 to 8.5]
  Week 20 | 8.4 [5.7 to 11.0] | 6.4 [4.0 to 8.8]
  Week 24 | 10.1 [7.1 to 13.0] | 7.5 [4.9 to 10.1]

14. Secondary Outcome: Part 1: Change From Baseline in Central Subfield Thickness in the Study Eye at Specified Timepoints Through Week 24
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the Bruch's membrane (BM) using optical coherence tomography (OCT), as assessed by the central reading center. The Mixed Model of Repeated Measures (MMRM) analysis included the categorical covariates of treatment arm, visit, visit-by-treatment arm interaction, baseline CST (continuous), and randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)] as fixed effects. An unstructured covariance structure was used. Missing data were implicitly imputed by MMRM model assuming missing at random. Treatment policy strategy (i.e., all observed values used) was applied to all intercurrent events (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
microns
  Week 4 | -420.8 [-429.2 to -412.5] | -417.3 [-425.6 to -409.0]
  Week 8 | -444.2 [-452.7 to -435.7] | -437.5 [-446.1 to -429.0]
  Week 12 | -451.0 [-460.6 to -441.5] | -442.5 [-452.1 to -433.0]
  Week 16 | -452.5 [-461.8 to -443.1] | -445.2 [-454.7 to -435.8]
  Week 20 | -459.4 [-467.8 to -451.0] | -445.1 [-453.6 to -436.6]
  Week 24 | -461.6 [-471.4 to -451.9] | -448.8 [-458.6 to -439.0]

15. Secondary Outcome: Part 1: Percentage of Participants With Absence of Macular Edema in the Study Eye at Specified Timepoints Through Week 24
Description: Absence of diabetic macular edema was defined as achieving a central subfield thickness of <325 microns in the study eye. Central subfield thickness was defined as the distance between the internal limiting membrane (ILM) and Bruch's membrane (BM) as assessed by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 83.8 [80.2 to 87.5] | 82.4 [78.5 to 86.2]
  Week 8 | 92.6 [90.0 to 95.2] | 91.2 [88.3 to 94.1]
  Week 12 | 93.4 [90.9 to 95.9] | 91.5 [88.6 to 94.3]
  Week 16 | 94.5 [92.2 to 96.8] | 92.8 [90.2 to 95.5]
  Week 20 | 94.8 [92.6 to 97.1] | 93.1 [90.5 to 95.7]
  Week 24 | 93.7 [91.2 to 96.2] | 92.0 [89.2 to 94.7]

16. Secondary Outcome: Part 1: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Intraretinal fluid was measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 45.5 [40.6 to 50.5] | 40.3 [35.6 to 45.0]
  Week 8 | 63.1 [58.3 to 68.0] | 61.7 [56.9 to 66.6]
  Week 12 | 53.2 [48.3 to 58.2] | 51.0 [46.2 to 55.9]
  Week 16 | 55.4 [50.5 to 60.3] | 51.9 [46.8 to 56.9]
  Week 20 | 59.0 [54.0 to 63.9] | 56.5 [51.6 to 61.5]
  Week 24 | 76.2 [71.9 to 80.5] | 70.8 [66.2 to 75.4]

17. Secondary Outcome: Part 1: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Subretinal fluid was measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 66.1 [61.4 to 70.8] | 65.0 [60.3 to 69.7]
  Week 8 | 89.6 [86.5 to 92.6] | 90.1 [87.0 to 93.1]
  Week 12 | 94.0 [91.6 to 96.4] | 93.9 [91.5 to 96.4]
  Week 16 | 95.3 [93.2 to 97.5] | 95.6 [93.5 to 97.7]
  Week 20 | 95.9 [93.9 to 97.9] | 94.5 [92.2 to 96.8]
  Week 24 | 96.4 [94.6 to 98.3] | 93.4 [90.8 to 95.9]

18. Secondary Outcome: Part 1: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 24
Description: Intraretinal fluid and subretinal fluid were measured in the study eye using optical coherence tomography (OCT) in the central subfield (center 1 mm) by a central reading center. The weighted percentage of participants was estimated based on the Cochran-Mantel Haenszel (CMH) weights stratified by randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)]. All observed values were used regardless of the occurrence of an intercurrent event (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). Missing assessments were imputed by last observation carried forward. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 33.0 [28.3 to 37.6] | 29.3 [24.9 to 33.7]
  Week 8 | 59.3 [54.4 to 64.1] | 59.3 [54.3 to 64.2]
  Week 12 | 52.7 [47.7 to 57.6] | 50.2 [45.3 to 55.1]
  Week 16 | 54.9 [49.9 to 59.8] | 51.3 [46.3 to 56.3]
  Week 20 | 58.2 [53.2 to 63.1] | 55.4 [50.5 to 60.4]
  Week 24 | 75.1 [70.8 to 79.5] | 68.6 [63.8 to 73.4]

19. Secondary Outcome: Part 1: Change From Baseline in National Eye Institute 25-Item Visual Functioning Questionnaire (NEI VFQ-25) Composite Score at Week 24
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and vision-related quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and 1 item on general health. The composite score ranges from 0 to 100, with higher scores indicating better vision-related functioning. For the ANCOVA analysis, the model uses the non-missing change from baseline in BCVA at Weeks 24 as the response variables adjusted for the treatment group, baseline NEI VFQ-25 Composite Score (continuous), baseline BCVA score (≥55 and ≤54 letters) and region (U.S. and Canada, Asia, and the rest of the world). Observed NEI VFQ-25 assessments were used regardless of the occurrence of intercurrent events. Missing data were not imputed. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Only participants with non-missing Baseline and Week 24 assessments were included for analysis.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1)
Number analyzed (Participants) | 339 | 330
score on a scale | 6.9 [5.8 to 8.0] | 8.1 [7.0 to 9.2]
Statistical Analysis 1: Comparison: Arm A: Faricimab Q4W (Part 1) vs Arm B: Aflibercept Q4W (Part 1); Test type: Other; Difference in Adjusted Means = -1.2, 95% CI 2-sided [-2.7 to 0.3], Standard Error of Mean 0.77

20. Secondary Outcome: Parts 1 and 2: Change From Baseline in BCVA in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
ETDRS Letters
  Week 4 | 13.6 [12.5 to 14.6] | 14.3 [13.3 to 15.4]
  Week 8 | 15.6 [14.4 to 16.8] | 16.5 [15.4 to 17.7]
  Week 12 | 17.0 [15.7 to 18.2] | 17.2 [15.9 to 18.4]
  Week 16 | 16.8 [15.5 to 18.1] | 17.6 [16.2 to 18.9]
  Week 20 | 17.0 [15.7 to 18.4] | 17.3 [15.9 to 18.6]
  Week 24 | 16.9 [15.5 to 18.3] | 17.3 [15.9 to 18.8]
  Week 28 | 16.0 [14.5 to 17.5] | 16.0 [14.4 to 17.5]
  Week 32 | 17.2 [15.7 to 18.7] | 17.5 [16.0 to 19.0]
  Week 36 | 17.0 [15.5 to 18.5] | 17.5 [15.9 to 19.0]
  Week 40 | 15.8 [14.2 to 17.5] | 16.2 [14.5 to 17.9]
  Week 44 | 16.5 [14.9 to 18.2] | 17.3 [15.7 to 19.0]
  Week 48 | 16.9 [15.2 to 18.5] | 17.6 [15.9 to 19.3]
  Week 52 | 16.4 [14.8 to 18.1] | 17.8 [16.2 to 19.5]
  Week 56 | 16.0 [14.3 to 17.7] | 16.9 [15.2 to 18.6]
  Week 60 | 16.9 [15.2 to 18.6] | 17.3 [15.6 to 19.0]
  Week 64 | 16.8 [15.1 to 18.5] | 17.2 [15.5 to 18.9]
  Week 68 | 16.9 [15.2 to 18.7] | 17.0 [15.2 to 18.7]
  Week 72 | 16.9 [15.1 to 18.6] | 17.1 [15.3 to 18.8]

21. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 41.5 [36.7 to 46.3] | 45.2 [40.4 to 49.9]
  Week 8 | 51.1 [46.3 to 55.9] | 53.7 [48.9 to 58.5]
  Week 12 | 54.6 [49.8 to 59.4] | 55.1 [50.3 to 59.9]
  Week 16 | 57.7 [52.8 to 62.5] | 59.5 [54.7 to 64.3]
  Week 20 | 56.6 [51.7 to 61.4] | 57.8 [53.0 to 62.6]
  Week 24 | 56.6 [51.7 to 61.5] | 58.1 [53.3 to 62.9]
  Week 28 | 53.3 [48.4 to 58.2] | 54.8 [50.0 to 59.6]
  Week 32 | 60.9 [56.1 to 65.8] | 57.6 [52.7 to 62.4]
  Week 36 | 58.2 [53.3 to 63.1] | 58.9 [54.2 to 63.7]
  Week 40 | 56.6 [51.7 to 61.4] | 55.9 [51.1 to 60.7]
  Week 44 | 55.7 [50.9 to 60.6] | 57.3 [52.5 to 62.1]
  Week 48 | 58.8 [53.9 to 63.6] | 58.1 [53.3 to 62.9]
  Week 52 | 57.6 [52.7 to 62.5] | 58.7 [53.8 to 63.5]
  Week 56 | 56.3 [51.3 to 61.2] | 57.3 [52.5 to 62.2]
  Week 60 | 58.2 [53.3 to 63.1] | 59.0 [54.1 to 63.8]
  Week 64 | 57.1 [52.3 to 61.9] | 59.5 [54.7 to 64.3]
  Week 68 | 56.8 [52.0 to 61.6] | 59.8 [54.9 to 64.6]
  Week 72 | 58.7 [53.9 to 63.6] | 60.0 [55.2 to 64.9]

22. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 60.9 [56.0 to 65.8] | 62.3 [57.6 to 66.9]
  Week 8 | 69.1 [64.5 to 73.7] | 72.8 [68.3 to 77.2]
  Week 12 | 73.2 [68.8 to 77.7] | 74.7 [70.3 to 79.0]
  Week 16 | 73.5 [69.1 to 78.0] | 75.8 [71.4 to 80.1]
  Week 20 | 72.4 [68.0 to 76.9] | 74.1 [69.7 to 78.5]
  Week 24 | 72.2 [67.7 to 76.6] | 73.3 [68.8 to 77.7]
  Week 28 | 69.7 [65.1 to 74.3] | 70.5 [66.0 to 75.1]
  Week 32 | 73.0 [68.5 to 77.4] | 74.4 [70.0 to 78.8]
  Week 36 | 73.8 [69.3 to 78.2] | 74.9 [70.6 to 79.3]
  Week 40 | 71.0 [66.5 to 75.6] | 73.0 [68.6 to 77.5]
  Week 44 | 71.6 [67.1 to 76.1] | 74.1 [69.7 to 78.5]
  Week 48 | 71.9 [67.3 to 76.4] | 75.5 [71.1 to 79.9]
  Week 52 | 71.0 [66.4 to 75.6] | 73.8 [69.4 to 78.3]
  Week 56 | 70.8 [66.2 to 75.3] | 72.2 [67.6 to 76.7]
  Week 60 | 72.7 [68.2 to 77.2] | 72.5 [67.9 to 77.0]
  Week 64 | 72.4 [67.9 to 76.9] | 71.6 [67.0 to 76.2]
  Week 68 | 72.1 [67.7 to 76.6] | 70.5 [65.9 to 75.1]
  Week 72 | 71.6 [67.1 to 76.1] | 73.0 [68.5 to 77.5]

23. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 83.1 [79.3 to 86.9] | 83.5 [79.7 to 87.2]
  Week 8 | 85.2 [81.7 to 88.8] | 86.8 [83.3 to 90.2]
  Week 12 | 87.4 [84.1 to 90.8] | 87.1 [83.7 to 90.5]
  Week 16 | 86.3 [82.9 to 89.8] | 88.7 [85.5 to 92.0]
  Week 20 | 84.1 [80.5 to 87.8] | 86.5 [83.0 to 90.0]
  Week 24 | 85.3 [81.8 to 88.8] | 84.6 [80.9 to 88.2]
  Week 28 | 81.7 [77.8 to 85.6] | 84.0 [80.3 to 87.7]
  Week 32 | 84.2 [80.5 to 87.8] | 87.3 [83.9 to 90.7]
  Week 36 | 84.7 [81.1 to 88.3] | 85.7 [82.1 to 89.3]
  Week 40 | 82.3 [78.4 to 86.1] | 84.3 [80.6 to 88.0]
  Week 44 | 82.8 [79.0 to 86.6] | 84.9 [81.2 to 88.5]
  Week 48 | 83.6 [79.9 to 87.3] | 83.7 [80.0 to 87.5]
  Week 52 | 80.9 [76.9 to 84.8] | 84.0 [80.3 to 87.8]
  Week 56 | 79.2 [75.2 to 83.3] | 81.5 [77.6 to 85.5]
  Week 60 | 82.8 [79.0 to 86.6] | 81.6 [77.6 to 85.5]
  Week 64 | 80.6 [76.6 to 84.6] | 81.5 [77.6 to 85.5]
  Week 68 | 83.3 [79.6 to 87.1] | 80.2 [76.1 to 84.2]
  Week 72 | 83.6 [79.9 to 87.3] | 79.6 [75.5 to 83.7]

24. Secondary Outcome: Parts 1 and 2: Percentage of Participants Gaining >0 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 92.1 [89.4 to 94.8] | 95.6 [93.5 to 97.7]
  Week 8 | 92.1 [89.4 to 94.8] | 94.8 [92.5 to 97.0]
  Week 12 | 93.2 [90.6 to 95.7] | 92.6 [89.9 to 95.2]
  Week 16 | 92.6 [90.0 to 95.3] | 92.0 [89.3 to 94.8]
  Week 20 | 90.5 [87.5 to 93.4] | 91.4 [88.6 to 94.3]
  Week 24 | 90.5 [87.5 to 93.4] | 89.2 [86.1 to 92.4]
  Week 28 | 88.0 [84.7 to 91.3] | 88.4 [85.2 to 91.7]
  Week 32 | 89.4 [86.2 to 92.5] | 92.0 [89.2 to 94.8]
  Week 36 | 89.9 [86.9 to 93.0] | 90.1 [87.0 to 93.1]
  Week 40 | 87.7 [84.5 to 91.0] | 88.7 [85.5 to 91.9]
  Week 44 | 88.5 [85.3 to 91.7] | 89.2 [86.1 to 92.4]
  Week 48 | 88.5 [85.3 to 91.7] | 88.7 [85.5 to 91.9]
  Week 52 | 85.8 [82.2 to 89.3] | 89.0 [85.8 to 92.2]
  Week 56 | 85.8 [82.3 to 89.3] | 87.3 [83.9 to 90.7]
  Week 60 | 86.6 [83.2 to 90.0] | 87.3 [83.9 to 90.7]
  Week 64 | 86.1 [82.6 to 89.6] | 86.2 [82.7 to 89.7]
  Week 68 | 87.4 [84.1 to 90.8] | 85.4 [81.8 to 89.0]
  Week 72 | 86.6 [83.2 to 90.1] | 85.7 [82.1 to 89.2]

25. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 98.4 [97.1 to 99.7] | 98.9 [97.8 to 100.0]
  Week 8 | 98.1 [96.7 to 99.5] | 98.1 [96.7 to 99.5]
  Week 12 | 98.6 [97.5 to 99.8] | 97.5 [95.9 to 99.1]
  Week 16 | 97.3 [95.6 to 98.9] | 97.0 [95.2 to 98.7]
  Week 20 | 97.0 [95.3 to 98.7] | 96.7 [94.9 to 98.5]
  Week 24 | 96.2 [94.3 to 98.1] | 96.7 [94.9 to 98.5]
  Week 28 | 95.6 [93.6 to 97.7] | 94.2 [91.8 to 96.6]
  Week 32 | 95.4 [93.3 to 97.5] | 96.1 [94.2 to 98.1]
  Week 36 | 95.4 [93.3 to 97.5] | 95.9 [93.8 to 97.9]
  Week 40 | 94.0 [91.6 to 96.4] | 95.9 [93.8 to 97.9]
  Week 44 | 94.0 [91.6 to 96.4] | 95.6 [93.5 to 97.7]
  Week 48 | 94.0 [91.6 to 96.4] | 95.6 [93.5 to 97.7]
  Week 52 | 94.6 [92.3 to 96.8] | 96.7 [94.9 to 98.5]
  Week 56 | 95.1 [92.9 to 97.3] | 95.6 [93.5 to 97.7]
  Week 60 | 93.5 [91.0 to 96.0] | 95.3 [93.2 to 97.5]
  Week 64 | 94.0 [91.6 to 96.4] | 94.8 [92.5 to 97.0]
  Week 68 | 93.5 [90.9 to 96.0] | 95.9 [93.8 to 97.9]
  Week 72 | 93.2 [90.6 to 95.7] | 95.0 [92.8 to 97.2]

26. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 98.1 [96.7 to 99.5] | 98.6 [97.4 to 99.8]
  Week 8 | 97.5 [96.0 to 99.1] | 97.5 [95.9 to 99.1]
  Week 12 | 97.8 [96.3 to 99.3] | 97.0 [95.2 to 98.7]
  Week 16 | 95.9 [93.9 to 97.9] | 96.1 [94.2 to 98.1]
  Week 20 | 96.7 [94.9 to 98.5] | 96.1 [94.2 to 98.1]
  Week 24 | 95.1 [92.9 to 97.3] | 95.9 [93.8 to 97.9]
  Week 28 | 94.6 [92.3 to 96.9] | 93.4 [90.9 to 95.9]
  Week 32 | 94.3 [91.9 to 96.6] | 95.9 [93.8 to 97.9]
  Week 36 | 94.3 [91.9 to 96.6] | 95.0 [92.8 to 97.3]
  Week 40 | 92.9 [90.3 to 95.5] | 93.9 [91.5 to 96.4]
  Week 44 | 93.2 [90.7 to 95.7] | 94.5 [92.2 to 96.8]
  Week 48 | 92.4 [89.7 to 95.0] | 93.9 [91.5 to 96.4]
  Week 52 | 92.9 [90.3 to 95.5] | 95.0 [92.8 to 97.2]
  Week 56 | 91.3 [88.4 to 94.1] | 93.6 [91.2 to 96.1]
  Week 60 | 92.1 [89.4 to 94.8] | 94.5 [92.2 to 96.8]
  Week 64 | 92.9 [90.3 to 95.5] | 93.9 [91.5 to 96.4]
  Week 68 | 92.6 [90.0 to 95.3] | 94.2 [91.8 to 96.6]
  Week 72 | 92.6 [90.0 to 95.3] | 93.7 [91.2 to 96.1]

27. Secondary Outcome: Parts 1 and 2: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Baseline in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 97.0 [95.3 to 98.7] | 98.1 [96.7 to 99.5]
  Week 8 | 96.2 [94.2 to 98.1] | 96.4 [94.5 to 98.3]
  Week 12 | 95.9 [93.9 to 97.9] | 96.1 [94.2 to 98.1]
  Week 16 | 95.4 [93.2 to 97.5] | 94.8 [92.5 to 97.0]
  Week 20 | 94.8 [92.6 to 97.1] | 93.9 [91.5 to 96.4]
  Week 24 | 94.0 [91.6 to 96.4] | 93.7 [91.2 to 96.1]
  Week 28 | 92.4 [89.7 to 95.1] | 91.7 [88.9 to 94.5]
  Week 32 | 91.3 [88.4 to 94.1] | 94.8 [92.5 to 97.0]
  Week 36 | 92.7 [90.0 to 95.3] | 94.2 [91.8 to 96.6]
  Week 40 | 91.0 [88.1 to 93.9] | 92.6 [89.9 to 95.2]
  Week 44 | 90.7 [87.8 to 93.6] | 92.8 [90.2 to 95.4]
  Week 48 | 91.0 [88.1 to 93.9] | 92.6 [89.9 to 95.2]
  Week 52 | 90.5 [87.5 to 93.4] | 93.4 [90.9 to 95.9]
  Week 56 | 88.5 [85.3 to 91.7] | 91.4 [88.6 to 94.3]
  Week 60 | 90.5 [87.5 to 93.4] | 92.3 [89.6 to 95.0]
  Week 64 | 90.7 [87.8 to 93.7] | 91.2 [88.3 to 94.1]
  Week 68 | 89.6 [86.6 to 92.7] | 91.7 [88.9 to 94.5]
  Week 72 | 90.5 [87.5 to 93.4] | 90.6 [87.7 to 93.6]

28. Secondary Outcome: Parts 1 and 2: Percentage of Participants Achieving ≥84 Letters in BCVA (20/20 Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 6.0 [3.6 to 8.4] | 4.7 [2.6 to 6.8]
  Week 8 | 8.7 [5.9 to 11.5] | 10.2 [7.2 to 13.2]
  Week 12 | 10.9 [7.8 to 14.0] | 11.9 [8.7 to 15.0]
  Week 16 | 11.5 [8.4 to 14.6] | 14.1 [10.7 to 17.5]
  Week 20 | 14.2 [10.9 to 17.6] | 14.9 [11.4 to 18.3]
  Week 24 | 14.5 [11.0 to 17.9] | 15.2 [11.7 to 18.7]
  Week 28 | 9.8 [6.9 to 12.8] | 12.7 [9.5 to 15.9]
  Week 32 | 13.4 [10.0 to 16.7] | 14.9 [11.4 to 18.3]
  Week 36 | 15.3 [11.8 to 18.8] | 14.9 [11.5 to 18.3]
  Week 40 | 14.8 [11.3 to 18.2] | 12.4 [9.2 to 15.7]
  Week 44 | 15.5 [12.0 to 19.1] | 14.1 [10.7 to 17.5]
  Week 48 | 15.0 [11.6 to 18.5] | 14.6 [11.2 to 18.0]
  Week 52 | 16.7 [13.0 to 20.3] | 14.9 [11.4 to 18.4]
  Week 56 | 14.8 [11.3 to 18.2] | 15.5 [12.0 to 18.9]
  Week 60 | 15.8 [12.3 to 19.4] | 16.3 [12.7 to 19.9]
  Week 64 | 16.1 [12.5 to 19.8] | 15.7 [12.2 to 19.3]
  Week 68 | 15.3 [11.8 to 18.9] | 15.2 [11.7 to 18.7]
  Week 72 | 15.3 [11.8 to 18.8] | 14.4 [11.0 to 17.7]

29. Secondary Outcome: Parts 1 and 2: Percentage of Participants Achieving ≥69 Letters in BCVA (20/40 or Better Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 45.0 [41.0 to 49.1] | 46.1 [41.9 to 50.2]
  Week 8 | 48.6 [44.3 to 52.8] | 54.6 [50.5 to 58.7]
  Week 12 | 54.9 [50.8 to 58.9] | 55.7 [51.4 to 60.0]
  Week 16 | 54.9 [50.6 to 59.1] | 59.3 [55.2 to 63.4]
  Week 20 | 54.1 [49.7 to 58.4] | 57.6 [53.4 to 61.8]
  Week 24 | 55.7 [51.3 to 60.0] | 59.0 [54.5 to 63.4]
  Week 28 | 53.2 [48.8 to 57.7] | 56.2 [51.8 to 60.7]
  Week 32 | 56.0 [51.6 to 60.4] | 60.4 [56.1 to 64.6]
  Week 36 | 53.8 [49.4 to 58.2] | 60.7 [56.3 to 65.0]
  Week 40 | 51.9 [47.3 to 56.4] | 56.2 [51.7 to 60.8]
  Week 44 | 53.0 [48.4 to 57.6] | 60.9 [56.5 to 65.3]
  Week 48 | 56.2 [51.8 to 60.7] | 60.6 [56.2 to 65.1]
  Week 52 | 54.3 [49.8 to 58.9] | 60.4 [55.9 to 64.8]
  Week 56 | 51.9 [47.3 to 56.4] | 58.7 [54.3 to 63.2]
  Week 60 | 56.0 [51.5 to 60.4] | 58.7 [54.3 to 63.1]
  Week 64 | 56.5 [52.1 to 61.0] | 57.9 [53.4 to 62.4]
  Week 68 | 56.0 [51.5 to 60.4] | 57.9 [53.4 to 62.4]
  Week 72 | 56.2 [51.7 to 60.8] | 58.5 [53.9 to 63.1]

30. Secondary Outcome: Parts 1 and 2: Percentage of Participants With ≤38 Letters in BCVA (20/200 or Worse Snellen Equivalent) in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 13
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 10.0 [7.3 to 12.8] | 8.6 [6.1 to 11.1]
  Week 8 | 8.2 [5.5 to 10.8] | 7.0 [4.6 to 9.4]
  Week 12 | 7.3 [4.9 to 9.8] | 6.4 [4.0 to 8.8]
  Week 16 | 7.8 [5.3 to 10.4] | 6.2 [3.8 to 8.5]
  Week 20 | 8.4 [5.7 to 11.0] | 6.4 [4.0 to 8.8]
  Week 24 | 10.1 [7.1 to 13.0] | 7.5 [4.9 to 10.1]
  Week 28 | 8.9 [6.1 to 11.7] | 9.4 [6.6 to 12.3]
  Week 32 | 9.2 [6.4 to 12.0] | 8.0 [5.4 to 10.7]
  Week 36 | 9.5 [6.6 to 12.4] | 8.3 [5.7 to 11.0]
  Week 40 | 9.8 [6.8 to 12.7] | 7.5 [4.9 to 10.1]
  Week 44 | 10.6 [7.5 to 13.6] | 8.3 [5.6 to 11.0]
  Week 48 | 10.0 [7.1 to 13.0] | 7.5 [4.9 to 10.1]
  Week 52 | 11.4 [8.3 to 14.5] | 7.2 [4.7 to 9.8]
  Week 56 | 11.9 [8.8 to 15.1] | 8.6 [5.8 to 11.4]
  Week 60 | 11.4 [8.3 to 14.5] | 8.3 [5.7 to 11.0]
  Week 64 | 11.1 [8.0 to 14.2] | 8.3 [5.6 to 11.0]
  Week 68 | 11.2 [8.0 to 14.3] | 8.3 [5.6 to 11.0]
  Week 72 | 11.4 [8.3 to 14.6] | 8.0 [5.4 to 10.7]

31. Secondary Outcome: Parts 1 and 2: Change From Baseline in NEI VFQ-25 Questionnaire Composite Score at Specified Timepoints Through Week 72
Description: The NEI VFQ-25 captures a patient's perception of vision-related functioning and vision-related quality of life. The core measure includes 25 items that comprise 11 vision-related subscales and 1 item on general health. The composite score ranges from 0 to 100, with higher scores indicating better vision-related functioning. For the MMRM analysis, the model adjusted for the treatment group, visit, visit-by-treatment group interaction, baseline NEI VFQ-25 Composite Score continuous), baseline BCVA score (≥55 and ≤54 letters), and region (U.S. and Canada, Asia, and the rest of the world). Observed NEI VFQ-25 assessments were used regardless of the occurrence of intercurrent events. Missing data were implicitly imputed. Invalid BCVA values were excluded. 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 24, 48, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
score on a scale
  Week 24 | 7.0 [5.9 to 8.0] | 8.2 [7.1 to 9.3]
  Week 48 | 7.0 [5.9 to 8.2] | 8.3 [7.1 to 9.5]
  Week 72 | 7.8 [6.5 to 9.0] | 8.5 [7.3 to 9.8]

32. Secondary Outcome: Parts 1 and 2: Change From Baseline in Central Subfield Thickness in the Study Eye at Specified Timepoints Through Week 72
Description: Central subfield thickness (CST) was defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) using optical coherence tomography (OCT), as assessed by the central reading center. The Mixed Model of Repeated Measures (MMRM) analysis included the categorical covariates of treatment arm, visit, visit-by-treatment arm interaction, baseline CST (continuous), and randomization stratification factors [baseline BCVA (≤34, 35-54, and ≥55 letters), and region (U.S. and Canada, Asia, and rest of the world)] as fixed effects. An unstructured covariance structure was used. Missing data were implicitly imputed by MMRM model assuming missing at random. Treatment policy strategy (i.e., all observed values used) was applied to all intercurrent events (discontinuation of treatment due to AEs or lack of efficacy, use of prohibited therapy). 95% CI is a rounding of 95.03% CI.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
microns
  Week 4 | -422.1 [-430.6 to -413.7] | -418.2 [-426.6 to -409.7]
  Week 8 | -445.1 [-453.6 to -436.6] | -438.5 [-447.0 to -429.9]
  Week 12 | -452.3 [-461.8 to -442.8] | -443.7 [-453.2 to -434.1]
  Week 16 | -453.8 [-463.1 to -444.5] | -446.2 [-455.5 to -436.9]
  Week 20 | -460.0 [-468.1 to -451.8] | -447.1 [-455.4 to -438.9]
  Week 24 | -462.3 [-472.3 to -452.3] | -447.8 [-457.9 to -437.8]
  Week 28 | -415.5 [-431.8 to -399.1] | -413.7 [-430.3 to -397.2]
  Week 32 | -459.4 [-468.7 to -450.1] | -445.8 [-455.3 to -436.3]
  Week 36 | -451.7 [-462.7 to -440.8] | -441.8 [-452.9 to -430.8]
  Week 40 | -409.8 [-425.6 to -394.0] | -414.0 [-429.9 to -398.0]
  Week 44 | -456.6 [-467.1 to -446.0] | -449.8 [-460.6 to -439.0]
  Week 48 | -461.2 [-471.3 to -451.1] | -448.0 [-458.3 to -437.7]
  Week 52 | -446.0 [-457.0 to -435.0] | -451.8 [-462.9 to -440.7]
  Week 56 | -435.9 [-449.8 to -422.0] | -426.2 [-440.3 to -412.1]
  Week 60 | -468.2 [-476.8 to -459.5] | -458.9 [-467.6 to -450.1]
  Week 64 | -466.6 [-473.7 to -459.5] | -465.5 [-472.6 to -458.3]
  Week 68 | -467.5 [-476.0 to -459.1] | -457.7 [-466.2 to -449.2]
  Week 72 | -463.5 [-472.8 to -454.3] | -458.6 [-467.9 to -449.2]

33. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Macular Edema in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 15
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 83.8 [80.2 to 87.5] | 82.4 [78.5 to 86.2]
  Week 8 | 92.6 [90.0 to 95.2] | 91.2 [88.3 to 94.1]
  Week 12 | 93.4 [90.9 to 95.9] | 91.5 [88.6 to 94.3]
  Week 16 | 94.5 [92.2 to 96.8] | 92.8 [90.2 to 95.5]
  Week 20 | 94.5 [92.2 to 96.8] | 93.1 [90.5 to 95.7]
  Week 24 | 93.7 [91.2 to 96.2] | 91.7 [88.9 to 94.5]
  Week 28 | 82.5 [78.6 to 86.4] | 84.0 [80.3 to 87.7]
  Week 32 | 93.2 [90.6 to 95.7] | 90.3 [87.4 to 93.3]
  Week 36 | 91.8 [89.0 to 94.6] | 89.5 [86.4 to 92.6]
  Week 40 | 80.0 [76.0 to 84.1] | 80.7 [76.7 to 84.7]
  Week 44 | 93.2 [90.6 to 95.7] | 90.9 [88.0 to 93.8]
  Week 48 | 92.6 [89.9 to 95.3] | 89.8 [86.7 to 92.9]
  Week 52 | 88.5 [85.2 to 91.8] | 90.9 [88.0 to 93.8]
  Week 56 | 87.4 [84.1 to 90.8] | 84.3 [80.6 to 88.0]
  Week 60 | 93.7 [91.3 to 96.2] | 92.8 [90.2 to 95.5]
  Week 64 | 94.3 [91.9 to 96.6] | 93.4 [90.8 to 95.9]
  Week 68 | 93.2 [90.6 to 95.7] | 91.4 [88.6 to 94.3]
  Week 72 | 92.4 [89.6 to 95.1] | 91.2 [88.3 to 94.0]

34. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Intraretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 16
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 45.5 [40.6 to 50.5] | 40.6 [35.8 to 45.3]
  Week 8 | 63.1 [58.3 to 68.0] | 61.7 [56.9 to 66.6]
  Week 12 | 53.2 [48.3 to 58.2] | 51.0 [46.2 to 55.9]
  Week 16 | 55.4 [50.5 to 60.3] | 51.9 [46.8 to 56.9]
  Week 20 | 59.0 [54.0 to 63.9] | 56.5 [51.6 to 61.5]
  Week 24 | 77.0 [72.8 to 81.3] | 70.8 [66.2 to 75.4]
  Week 28 | 53.8 [48.7 to 58.9] | 51.5 [46.4 to 56.6]
  Week 32 | 67.7 [63.1 to 72.4] | 67.2 [62.5 to 72.0]
  Week 36 | 62.8 [58.1 to 67.5] | 57.6 [52.6 to 62.6]
  Week 40 | 52.7 [47.7 to 57.7] | 51.0 [46.0 to 56.1]
  Week 44 | 66.4 [61.6 to 71.2] | 63.4 [58.5 to 68.3]
  Week 48 | 74.3 [69.9 to 78.8] | 69.7 [65.0 to 74.3]
  Week 52 | 66.9 [62.2 to 71.6] | 63.4 [58.5 to 68.2]
  Week 56 | 60.9 [56.0 to 65.9] | 58.7 [53.7 to 63.6]
  Week 60 | 71.6 [67.0 to 76.1] | 72.7 [68.2 to 77.2]
  Week 64 | 76.5 [72.2 to 80.8] | 72.7 [68.2 to 77.2]
  Week 68 | 74.6 [70.2 to 79.0] | 71.3 [66.8 to 75.9]
  Week 72 | 78.1 [73.9 to 82.3] | 74.4 [69.9 to 78.9]

35. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 17
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 66.1 [61.4 to 70.8] | 65.0 [60.3 to 69.7]
  Week 8 | 89.6 [86.5 to 92.6] | 90.1 [87.0 to 93.1]
  Week 12 | 94.0 [91.6 to 96.4] | 93.9 [91.5 to 96.4]
  Week 16 | 95.3 [93.2 to 97.5] | 95.6 [93.5 to 97.7]
  Week 20 | 95.9 [93.9 to 97.9] | 94.5 [92.2 to 96.8]
  Week 24 | 96.2 [94.2 to 98.1] | 93.4 [90.8 to 95.9]
  Week 28 | 89.3 [86.2 to 92.5] | 90.1 [87.0 to 93.1]
  Week 32 | 95.6 [93.6 to 97.7] | 94.5 [92.2 to 96.8]
  Week 36 | 95.1 [92.9 to 97.3] | 92.3 [89.6 to 95.0]
  Week 40 | 89.6 [86.5 to 92.7] | 89.3 [86.1 to 92.4]
  Week 44 | 95.4 [93.2 to 97.5] | 92.8 [90.2 to 95.5]
  Week 48 | 93.4 [90.9 to 95.9] | 89.5 [86.4 to 92.6]
  Week 52 | 92.6 [89.9 to 95.3] | 93.6 [91.2 to 96.1]
  Week 56 | 93.4 [90.9 to 95.9] | 90.1 [87.1 to 93.1]
  Week 60 | 97.0 [95.3 to 98.7] | 94.8 [92.5 to 97.0]
  Week 64 | 96.7 [94.9 to 98.5] | 95.9 [93.8 to 97.9]
  Week 68 | 97.6 [96.0 to 99.1] | 93.9 [91.6 to 96.3]
  Week 72 | 95.4 [93.2 to 97.5] | 93.1 [90.6 to 95.7]

36. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Absence of Intraretinal Fluid and Subretinal Fluid in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 18
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 4 | 33.0 [28.3 to 37.6] | 29.3 [24.9 to 33.7]
  Week 8 | 59.3 [54.4 to 64.1] | 59.3 [54.3 to 64.2]
  Week 12 | 52.7 [47.7 to 57.6] | 50.2 [45.3 to 55.1]
  Week 16 | 54.9 [49.9 to 59.8] | 51.3 [46.3 to 56.3]
  Week 20 | 58.2 [53.2 to 63.1] | 55.4 [50.5 to 60.4]
  Week 24 | 76.0 [71.6 to 80.3] | 68.6 [63.8 to 73.4]
  Week 28 | 52.7 [47.6 to 57.8] | 51.2 [46.1 to 56.3]
  Week 32 | 67.2 [62.6 to 71.8] | 66.4 [61.6 to 71.2]
  Week 36 | 62.8 [58.1 to 67.5] | 56.5 [51.5 to 61.5]
  Week 40 | 52.7 [47.7 to 57.7] | 50.2 [45.1 to 55.2]
  Week 44 | 64.7 [59.9 to 69.6] | 60.9 [56.0 to 65.8]
  Week 48 | 70.8 [66.1 to 75.4] | 65.8 [61.0 to 70.6]
  Week 52 | 65.8 [61.1 to 70.6] | 61.7 [56.8 to 66.6]
  Week 56 | 60.7 [55.7 to 65.6] | 58.1 [53.2 to 63.0]
  Week 60 | 71.0 [66.4 to 75.6] | 71.6 [67.0 to 76.2]
  Week 64 | 75.4 [71.1 to 79.8] | 71.9 [67.3 to 76.4]
  Week 68 | 74.3 [69.9 to 78.8] | 70.8 [66.2 to 75.3]
  Week 72 | 77.0 [72.8 to 81.3] | 71.6 [67.0 to 76.3]

37. Secondary Outcome: Part 2: Change From Week 24 in BCVA in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 1
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: Intent-to-Treat (ITT) Population: all participants who were randomized in the study, grouped according to the treatment assigned at randomization. Participants with evaluable Week 24 BCVA were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: ETDRS Letters
Groups:
- Arm A: Faricimab Q4W to Faricimab PTI (Part 2): In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
- Arm B: Aflibercept Q4W to Faricimab PTI (Part 2): In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was to be administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 340 | 331
ETDRS Letters
  Week 28 | -0.8 [-1.6 to 0.0] | -1.2 [-2.0 to -0.4]
  Week 32 | 0.2 [-0.6 to 0.9] | 0.2 [-0.6 to 1.0]
  Week 36 | -0.1 [-0.8 to 0.7] | 0.1 [-0.7 to 0.9]
  Week 40 | -1.3 [-2.4 to -0.2] | -1.4 [-2.4 to -0.3]
  Week 44 | -0.6 [-1.6 to 0.4] | 0.0 [-1.0 to 1.0]
  Week 48 | -0.1 [-1.1 to 0.9] | 0.2 [-0.8 to 1.1]
  Week 52 | -0.6 [-1.6 to 0.4] | 0.3 [-0.6 to 1.3]
  Week 56 | -1.1 [-2.1 to 0.0] | -0.6 [-1.7 to 0.5]
  Week 60 | 0.0 [-1.1 to 1.0] | -0.1 [-1.2 to 0.9]
  Week 64 | -0.2 [-1.3 to 0.8] | -0.2 [-1.3 to 0.9]
  Week 68 | -0.1 [-1.2 to 1.0] | -0.5 [-1.6 to 0.6]
  Week 72 | -0.2 [-1.3 to 1.0] | -0.3 [-1.5 to 0.8]

38. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 28 | 86.3 [82.9 to 89.8] | 83.8 [80.0 to 87.5]
  Week 32 | 88.8 [85.6 to 92.0] | 87.9 [84.6 to 91.2]
  Week 36 | 89.3 [86.2 to 92.5] | 87.9 [84.6 to 91.2]
  Week 40 | 87.4 [84.0 to 90.8] | 86.0 [82.4 to 89.5]
  Week 44 | 87.4 [84.0 to 90.8] | 88.4 [85.2 to 91.7]
  Week 48 | 88.5 [85.3 to 91.7] | 87.3 [83.9 to 90.7]
  Week 52 | 86.3 [82.8 to 89.8] | 87.6 [84.2 to 91.0]
  Week 56 | 85.7 [82.2 to 89.3] | 85.4 [81.8 to 89.0]
  Week 60 | 87.7 [84.3 to 91.0] | 86.2 [82.7 to 89.8]
  Week 64 | 86.3 [82.8 to 89.8] | 85.9 [82.4 to 89.5]
  Week 68 | 87.1 [83.7 to 90.5] | 85.4 [81.8 to 89.0]
  Week 72 | 86.6 [83.1 to 90.0] | 84.0 [80.3 to 87.8]

39. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥10 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 28 | 82.8 [79.0 to 86.6] | 81.3 [77.3 to 85.2]
  Week 32 | 87.1 [83.7 to 90.6] | 86.0 [82.4 to 89.5]
  Week 36 | 84.7 [81.0 to 88.4] | 85.4 [81.8 to 89.0]
  Week 40 | 82.8 [78.9 to 86.6] | 81.6 [77.6 to 85.5]
  Week 44 | 84.1 [80.4 to 87.9] | 86.8 [83.4 to 90.2]
  Week 48 | 84.4 [80.7 to 88.1] | 84.8 [81.2 to 88.5]
  Week 52 | 82.8 [78.9 to 86.6] | 85.4 [81.8 to 89.0]
  Week 56 | 80.0 [76.0 to 84.1] | 81.8 [77.9 to 85.8]
  Week 60 | 83.6 [79.8 to 87.4] | 82.6 [78.8 to 86.5]
  Week 64 | 81.7 [77.7 to 85.6] | 83.2 [79.4 to 87.0]
  Week 68 | 82.2 [78.3 to 86.1] | 80.7 [76.7 to 84.7]
  Week 72 | 82.5 [78.6 to 86.3] | 80.7 [76.7 to 84.7]

40. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of ≥5 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 28 | 72.7 [68.2 to 77.2] | 69.7 [65.0 to 74.4]
  Week 32 | 78.4 [74.2 to 82.6] | 75.5 [71.1 to 79.9]
  Week 36 | 74.1 [69.6 to 78.5] | 80.2 [76.1 to 84.2]
  Week 40 | 71.0 [66.4 to 75.6] | 71.6 [67.0 to 76.2]
  Week 44 | 73.7 [69.3 to 78.2] | 73.0 [68.5 to 77.6]
  Week 48 | 76.5 [72.2 to 80.8] | 74.1 [69.6 to 78.6]
  Week 52 | 71.3 [66.7 to 75.9] | 74.1 [69.6 to 78.6]
  Week 56 | 69.4 [64.7 to 74.1] | 68.3 [63.6 to 73.1]
  Week 60 | 74.3 [69.8 to 78.7] | 71.6 [67.0 to 76.2]
  Week 64 | 74.6 [70.1 to 79.0] | 71.6 [67.0 to 76.2]
  Week 68 | 73.2 [68.7 to 77.7] | 69.2 [64.5 to 73.8]
  Week 72 | 72.9 [68.4 to 77.5] | 70.3 [65.6 to 74.9]

41. Secondary Outcome: Part 2: Percentage of Participants Avoiding a Loss of >0 Letters in BCVA From Week 24 in the Study Eye at Specified Timepoints Through Week 72
Description: as for outcome 3
Time Frame: Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, and 72
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 366 | 363
Percentage of participants
  Week 28 | 48.9 [43.8 to 54.0] | 45.4 [40.4 to 50.5]
  Week 32 | 56.0 [50.9 to 61.1] | 52.9 [47.8 to 58.0]
  Week 36 | 55.5 [50.4 to 60.5] | 55.1 [50.0 to 60.2]
  Week 40 | 53.0 [47.9 to 58.0] | 48.2 [43.1 to 53.3]
  Week 44 | 53.0 [47.9 to 58.0] | 54.0 [49.0 to 59.1]
  Week 48 | 56.5 [51.5 to 61.6] | 53.5 [48.4 to 58.6]
  Week 52 | 56.0 [50.9 to 61.1] | 56.5 [51.4 to 61.5]
  Week 56 | 54.9 [49.8 to 60.0] | 53.2 [48.1 to 58.2]
  Week 60 | 55.9 [50.9 to 61.0] | 51.0 [45.9 to 56.1]
  Week 64 | 54.6 [49.5 to 59.7] | 52.1 [47.0 to 57.2]
  Week 68 | 55.4 [50.4 to 60.4] | 52.3 [47.3 to 57.4]
  Week 72 | 55.4 [50.4 to 60.5] | 52.7 [47.6 to 57.7]

42. Secondary Outcome: Part 2: Percentage of Participants on Different Treatment Intervals at Week 68
Description: In Part 2 of the study, participants in both the faricimab Q4W and aflibercept Q4W arms in Part 1 received 6 mg faricimab intravitreal injections administered according to a personalized treatment interval (PTI) dosing regimen in intervals between Q4W and Q16W. At faricimab dosing visits, treatment intervals were maintained or adjusted (i.e., increased by 4 weeks or decreased by 4, 8, or 12 weeks), based on central subfield thickness (CST) and BCVA values.
Time Frame: Week 68
Population: The analysis population included all randomized participants who had not discontinued the study at Week 68 and with available treatment interval information.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 330 | 315
Percentage of participants
  Once Every 4 Weeks (Q4W) | 34.5 [29.4 to 39.7] | 32.4 [27.2 to 37.6]
  Once Every 8 Weeks (Q8W) | 20.0 [15.7 to 24.3] | 17.5 [13.3 to 21.7]
  Once Every 12 Weeks (Q12W) | 8.5 [5.5 to 11.5] | 11.1 [7.6 to 14.6]
  Once Every 16 Weeks (Q16W) | 37.0 [31.8 to 42.2] | 39.0 [33.7 to 44.4]

43. Secondary Outcome: Part 2: Number of Study Drug Injections Received in the Study Eye From Week 24 Through Week 72
Time Frame: From Week 24 to Week 72
Population: Safety-Evaluable Population: All participants randomized in the study who received at least one injection of active study drug in the study eye. For Part 2, the safety analysis included: in Arm A, all participants with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168; in Arm B, all participants who received at least one faricimab dose.
Measure: Median (Full Range); unit: Injections
Arm/Group | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 359 | 342
Injections | 5.0 [1 to 12] | 4.0 [1 to 12]

44. Secondary Outcome: Incidence and Severity of Ocular Adverse Events in the Study Eye, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This analysis of adverse events (AEs) only includes ocular AEs that occurred in the study eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: Safety-Evaluable Population: All participants randomized in the study who received at least one injection of active study drug (faricimab or aflibercept) in the study eye. For Part 2, the safety analysis included: in Arm A, all participants with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168; in Arm B, all participants who received at least one faricimab dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 365 | 361 | 359 | 342
Participants
  Adverse Event (AE) | 89 | 98 | 130 | 118
  AE by Severity: Mild | 65 | 65 | 63 | 69
  AE by Severity: Moderate | 18 | 27 | 52 | 43
  AE by Severity: Severe | 6 | 6 | 15 | 6
  Serious Adverse Event (SAE) | 9 | 13 | 26 | 12
  AE Leading to Withdrawal from Study Treatment | 3 | 2 | 5 | 3
  Treatment Related AEs | 15 | 6 | 14 | 11
  Treatment Related SAEs | 3 | 2 | 4 | 0
  Any AE of Special Interest (AESI) | 8 | 12 | 21 | 9
  AESI: Drop in Visual Acuity Score ≥30 | 6 | 6 | 15 | 7
  AESI: Associated with Severe IOI | 0 | 0 | 0 | 1
  AESI: Intervention Req. to Prevent Permanent Vision Loss | 2 | 6 | 6 | 1

45. Secondary Outcome: Incidence of Ocular Adverse Events in the Fellow Eye
Description: This analysis of adverse events (AEs) only includes ocular AEs that occurred in the fellow eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. Ocular AEs of special interest included the following: Suspected transmission of an infectious agent by the study drug; Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, require surgical or medical intervention to prevent permanent loss of sight, or are associated with severe intraocular inflammation (IOI).
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 365 | 361 | 359 | 342
Participants
  Adverse Event (AE) | 31 | 33 | 70 | 51
  Serious Adverse Event (SAE) | 1 | 1 | 1 | 0
  Any AE of Special Interest (AESI) | 1 | 1 | 1 | 0
  AESI: Drop in Visual Acuity Score ≥30 | 1 | 1 | 1 | 0

46. Secondary Outcome: Incidence of Non-Ocular Adverse Events
Description: This analysis of adverse events (AEs) only includes non-ocular (systemic) AEs. Investigators sought information on adverse events (AEs) at each contact with the participants. All AEs were recorded and the investigator made an assessment of seriousness, severity, and causality of each AE. The non-ocular AE of special interest was: Cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
Number analyzed (Participants) | 365 | 361 | 359 | 342
Participants
  Adverse Event (AE) | 123 | 134 | 191 | 174
  Serious Adverse Event (SAE) | 22 | 23 | 30 | 41
  AE Leading to Withdrawal from Study Treatment | 0 | 1 | 3 | 3
  Any AE of Special Interest (AESI) | 0 | 0 | 0 | 0

47. Secondary Outcome: Plasma Concentration of Faricimab Over Time
Time Frame: Predose at Day 1 (Baseline), Weeks 4, 24, 28, 52, and 72
Population: Pharmacokinetic-Evaluable Population: All safety-evaluable participants randomized to faricimab arm or who received faricimab with at least one plasma sample, provided sufficient dosing information (dose and dosing time) was available. The number analyzed indicates all participants who provided a PK sample at a given timepoint.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (μg/mL)
Groups:
- Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2): In Part 1 (Day 1 through Week 24), participants were randomly assigned to Arm A to receive faricimab 6 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
- Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2): In Part 1 (Day 1 through Week 24), participants were randomly assigned to Arm B to receive aflibercept 2 milligrams (mg) by IVT injection once every 4 weeks (Q4W) from Day 1 through Week 20 (a total of 6 injections). In Part 2 (from Week 24 to Week 72), participants received faricimab 6 mg by IVT injection according to a personalized treatment interval (PTI) dosing regimen. To preserve masking for Part 2, a sham procedure was to be administered during study visits at which no faricimab treatment was administered (according to the PTI dosing regimen).
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2)
Number analyzed (Participants) | 365 | 342
microgram per millilitre (μg/mL)
  Baseline: number analyzed (Participants) | 359 | 0
  Baseline | 0.0001 (0.0009) |
  Week 4: number analyzed (Participants) | 345 | 0
  Week 4 | 0.0222 (0.0176) |
  Week 24: number analyzed (Participants) | 321 | 324
  Week 24 | 0.0257 (0.0217) | 0.0005 (0.0014)
  Week 28: number analyzed (Participants) | 323 | 314
  Week 28 | 0.0055 (0.0086) | 0.0026 (0.0084)
  Week 52: number analyzed (Participants) | 318 | 300
  Week 52 | 0.0089 (0.0142) | 0.0090 (0.0136)
  Week 72: number analyzed (Participants) | 279 | 272
  Week 72 | 0.0087 (0.0140) | 0.0099 (0.0167)

48. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Faricimab at Baseline and Post-Baseline During the Study
Description: Anti-drug antibodies (ADAs) against fariciamb were detected in plasma using a validated bridging enzyme-linked immunosorbent assay (ELISA). The number of participants with treatment-emergent ADA-positive samples includes post-baseline evaluable participants with at least one treatment-induced (defined as having an ADA-negative sample or missing sample at baseline and any positive post-baseline sample) or treatment-boosted (defined as having an ADA-positive sample at baseline and any positive post-baseline sample with a titer that is equal to or greater than 4-fold baseline titer) ADA-positive sample during the study treatment period. Treatment-unaffected ADA-positive is a post-baseline sample with a titer that is lower than 4-fold the ADA-positive baseline titer (faricimab arm) or the ADA-positive titer prior to first faricimab injection (aflibercept arm).
Time Frame: Predose at Day 1 (Baseline), Weeks 4, 24, 28, 52, and 72
Population: The immunogenicity analysis included all participants with an evaluable ADA sample. At baseline, evaluable participants were those with an ADA sample prior to faricimab injection, including those who did not receive study treatment; post-baseline, evaluable participants were those with an ADA sample after having received at least one dose of faricimab.
Measure: Count of Participants; unit: Participants
Groups:
- All Faricimab Participants: This immunogenicity analysis group represents all participants with an evaluable ADA sample. At baseline, evaluable participants were those with an ADA sample prior to faricimab injection, including those who did not receive study treatment; post-baseline, evaluable participants were those with an ADA sample after having received at least one dose of faricimab.
Arm/Group | Arm A: Faricimab Q4W (Part 1), Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W (Part 1), Faricimab PTI (Part 2) | All Faricimab Participants
Number analyzed (Participants) | 366 | 342 | 708
Participants
  Baseline (BL): Total ADA-Positive: number analyzed (Participants) | 362 | 342 | 704
  Baseline (BL): Total ADA-Positive | 4 | 5 | 9
  Post-BL: Total ADA-Positive: number analyzed (Participants) | 364 | 342 | 706
  Post-BL: Total ADA-Positive | 62 | 27 | 89
  Post-BL: Treatment-Emergent ADA-Positive: number analyzed (Participants) | 364 | 342 | 706
  Post-BL: Treatment-Emergent ADA-Positive | 60 | 23 | 83
  Post-BL: Treatment-Unaffected ADA-Positive: number analyzed (Participants) | 364 | 342 | 706
  Post-BL: Treatment-Unaffected ADA-Positive | 2 | 4 | 6

ADVERSE EVENTS:
Time Frame: Part 1: From first dose up to Week 24; Part 2: from Week 24 through Week 72
Description: Adverse events (AEs) are reported for the safety population, which includes all participants who received ≥1 injection of active study drug (faricimab or aflibercept) in the study eye. For Part 2, safety analysis included: in Arm A, those with Week 24 treatment or dose hold, or if none, follow-up beyond Day 168; in Arm B, those who received ≥1 faricimab dose. For ocular AEs, the number of participants and events reported per term are specified to have occurred in the study eye or the fellow eye.
Arm/Group | Arm A: Faricimab Q4W (Part 1) | Arm B: Aflibercept Q4W (Part 1) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2)
All-Cause Mortality (participants affected / at risk) | 1/365 | 2/361 | 4/359 | 1/342
Serious Adverse Events (participants affected / at risk) | 32/365 | 34/361 | 55/359 | 51/342
Other Adverse Events (participants affected / at risk) | 67/365 | 66/361 | 109/359 | 118/342
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab Q4W (Part 1) (N=365) | Arm B: Aflibercept Q4W (Part 1) (N=361) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) (N=359) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2) (N=342)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — AEs occurred in the fellow eye
Cystoid macular oedema (Eye disorders) | 2 (2) | 2 (2) | 5 (6) | 1 (1) — AEs occurred in the study eye
Macular ischaemia (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) — AEs occurred in the study eye
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — AEs occurred in the study eye
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — AEs occurred in the study eye
Retinal artery occlusion (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) — AEs occurred in the study eye
Retinal ischaemia (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) — AEs occurred in the study eye
Retinal tear (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) — AEs occurred in the study eye
Retinal vein occlusion (Eye disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3) — AEs occurred in the study eye
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — AEs occurred in the study eye
Uveitis (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Duodenal bulb deformity (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — AEs occurred in the study eye
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — AEs occurred in the study eye
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — AEs occurred in the study eye
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — AEs occurred in the fellow eye
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mesenteric lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the fellow eye
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AEs occurred in the study eye
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Iris neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AEs occurred in the study eye
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — AEs occurred in the study eye
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — AEs occurred in the study eye
Vitritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — AEs occurred in the study eye
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stent-graft endoleak (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secondary hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — AEs occurred in the study eye
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Faricimab Q4W (Part 1) (N=365) | Arm B: Aflibercept Q4W (Part 1) (N=361) | Arm A: Faricimab Q4W to Faricimab PTI (Part 2) (N=359) | Arm B: Aflibercept Q4W to Faricimab PTI (Part 2) (N=342)
Conjunctival haemorrhage (Eye disorders) | 10 (11) | 14 (14) | 10 (11) | 7 (8) — AEs occurred in the study eye
Vitreous detachment (Eye disorders) | 11 (11) | 9 (9) | 6 (6) | 14 (14) — AEs occurred in the study eye
COVID-19 (Infections and infestations) | 14 (14) | 12 (12) | 42 (42) | 46 (46)
Intraocular pressure increased (Investigations) | 9 (11) | 12 (22) | 16 (21) | 15 (34) — AEs occurred in the study eye
Hypertension (Vascular disorders) | 15 (15) | 10 (10) | 12 (13) | 8 (8)
Cataract (Eye disorders) | 3 (3) | 7 (7) | 14 (14) | 14 (14) — AEs occurred in the study eye
Cystoid macular oedema (Eye disorders) | 1 (1) | 3 (3) | 11 (15) | 10 (10) — AEs occurred in the study eye
Macular oedema (Eye disorders) | 2 (2) | 0 (0) | 7 (12) | 14 (16) — AEs occurred in the study eye
Epiretinal membrane (Eye disorders) | 3 (3) | 2 (2) | 3 (3) | 11 (11) — AEs occurred in the study eye
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (7) | 10 (10) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04740931/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04740931/SAP_001.pdf